CLINICAL TRIAL: NCT05625451
Title: A Comparison Between Two Intervals of Daily Total End Range Time for Treatment of Proximal Interphalangeal Joint Flexion Contracture Using an Elastic Tension Digital Neoprene Orthosis
Brief Title: High Doses of Total End Range Time Offer Better Results Than Low Doses Treating Proximal Interphalangeal Joint Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vicenç Punsola Izard (Other)
Responsible Party: Sponsor-Investigator, Vicenç Punsola Izard, Physical Therapist, Certified Hand Therapist in Hand Therapy Barcelona, MSc Gimbernat Universiy , Assistant lecturer at Gimbernat University, PhD Candidate at University of Barcelona, Hand Therapy Barcelona
Organization: Hand Therapy Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2022-11-07; First posted 2022-11-23 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Proximal Interphalangeal Finger Joint Contractures

STUDY DESIGN:
Intervention Model Description: Randomized parallel-group trial with concealed allocation, assessor blinding and intention-to-treat
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20-22 hours of daily total end range time intervention (Experimental): used the elastic tension digital neoprene orthosis from twenty to twenty-two hours
  Interventions: Device: Elastic Tension Digital Neoprene Orthosis
- 11-13 hours daily total end range time intervention (Active Comparator): used the elastic tension digital neoprene orthosis from eleven to thirteen hours
  Interventions: Device: Elastic Tension Digital Neoprene Orthosis

INTERVENTIONS:
Device: Elastic Tension Digital Neoprene Orthosis — The treatment consisted of an exercise program in conjunction with the use of an extension elastic tension digital neoprene orthosis to generate two different daily total end range time doses. Group A patients used a dose of twenty to twenty-two hours of daily total end range time while group B patients used the extension elastic tension digital neoprene orthosis to achieve a daily total end range time between eleven and thirteen hours for a mean of twenty hours a day. The exercise program was the same for both groups.

SUMMARY:
Elastic Tension Digital Neoprene Orthosis is a new device that can increase the dose of treatment of the proximal interphalangeal flexion contractures. This treatment improved the results in extension and also reducing the time to obtain it.

DETAILED DESCRIPTION:
Question: In fingers with proximal interphalangeal joint flexion contractures, do significant differences exist between the passive range of motion improvement achieved in joints that receive higher doses of daily total end range time compared to those that receive lower doses of daily total end range time?

Design: Randomized parallel-group trial with concealed allocation, assessor blinding and intention-to-treat

Participants: Fifty-seven fingers in fifty patients suffering a proximal interphalangeal joint flexion contracture

Intervention: The treatment consisted of an exercise program in conjunction with the use of an extension elastic tension digital neoprene orthosis to generate extension. Researchers applied two different daily total end range time doses. Group A patients used the orthosis with a dose of twenty to twenty-two hours of daily total end range time while group B patients used the elastic tension digital neoprene orthosis to achieve a daily total end range time between eleven and thirteen hours. The exercise program was the same for both groups.

Outcome measures: The researchers performed the goniometric measurements manually twice at the beginning of every session during the three-week period. The first measurement was at the patient arrival after a preconditioning and the second was after twenty minutes. This measurement at the first session was included as a Modified weeks test while at the second, third and forth session was recorded as a contraction test. Patient report of orthosis wear time and

ELIGIBILITY:
Patient Inclusion Criteria:

* Patients with flexion contractures of the proximal interphalangeal joint after trauma or post-surgical complications.
* Patients with long standing flexion contractures
* Patients with contractures greater than 45º.

Exclusion Criteria:

* Patients with acute tendon injuries or fractures
* Patients with inflammatory conditions,
* Patients with proximal interphalangeal joint replacements,
* Patients with Dupuytren conservative treatments
* Patients lacking active proximal interphalangeal joint extension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Change in the proximal interphalangeal joint extension | 7 days
  difference in passive finger extension between the first day and the seventh day
Change in the proximal interphalangeal joint extension | 21 days
  difference in passive finger extension between the first day and the twenty first day
- Modified Weeks Test | fifteen minutes
  Difference in finger extension at the beginning of te session and after a 15 min passive assisted extension exercise with a force of 500g
- Contraction Test | 21 days
  Finger reaction at release of the orthosis

CONTACTS AND LOCATIONS:
Locations (1):
- Hand Therapy Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No